CLINICAL TRIAL: NCT06374342
Title: Safety and Clinical Performance Assessment of Bone Substitutes Used for Bone Voids Filling - A Post-Market Clinical Follow-Up
Brief Title: Bone Substitutes Outcomes - Post Market Follow-up
Status: Recruiting | Type: Observational
Sponsor: Teknimed (Industry)
Responsible Party: Sponsor
Other Study IDs: SO01-TK-SUBSTITUTES
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Bone Resorption
Keywords: Bone substitutes; Gel; Hydroxyapatite; Tricalcium phosphate; Calcium phosphate; Ceramics
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (8):
- CERAFORM Granules Orthopedics: Bone grafting
  Interventions: Device: Bone defect
- CERAFORM Granules Spine: Spinal fusion
  Interventions: Device: Spine fusion
- CERAFORM Sticks Orthopedics: Bone grafting
  Interventions: Device: Bone defect
- CERAFORM Wedge Orthopedics: Bone grafting
  Interventions: Device: Bone defect
- TRIHA+ Spine: Spinal fusion
  Interventions: Device: Spine fusion
- TRIHA+ Orthopedics: Bone grafting
  Interventions: Device: Bone defect
- NANOGEL Spine: Cage filling
  Interventions: Device: Cage filling
- NANOGEL Orthopedics: Bone grafting
  Interventions: Device: Bone defect

INTERVENTIONS:
Device: Bone defect — Bone grafting is a procedure where damaged bones can be repaired or rebuilt using transplanted bone from another source. Sources for transplant bone include the patient (autograft), a cadaver (allograft) or synthetic bone.
  Groups: CERAFORM Granules Orthopedics; CERAFORM Sticks Orthopedics; CERAFORM Wedge Orthopedics; NANOGEL Orthopedics; TRIHA+ Orthopedics
Device: Spine fusion — Spinal fusion is a surgery procedure that reinforces your back structure and stability by linking two vertebrae together
  Groups: CERAFORM Granules Spine; TRIHA+ Spine
Device: Cage filling — Intervertebral fusion with cages is a surgical procedure used to stabilize the spine by fusing adjacent vertebrae. The cages, typically made of materials like titanium or plastic, and pre-filled with bone graft substitutes are placed between the vertebrae to maintain the proper spacing and alignment.
  Groups: NANOGEL Spine

SUMMARY:
A Post-Market Clinical Follow-Up (PMCF) Study to collect clinical data on safety and performance of all TEKNIMED Bone Substitute range of products: CERAFORM, TRIHA+, NANOGEL, and all their private labels.

TEKNIMED bone substitutes are legacy products, some marketed for more than 20 years. Their performance and safety have already been demonstrated by Post-Market Surveillance and previous clinical studies. The current Post-Market Clinical Follow-Up study aims to confirm these claims by collecting data in a "real-life" setting.

The study is a retrospective and prospective global, single arm, non-controlled, multicentric, prospective observational study. Patients will be followed as per local standard medical care of the sites.

DETAILED DESCRIPTION:
It is admitted that:

* Surgeons are often concerned by bone void filling and they can choose between synthetic bone substitutes or bone grafts of animal or human origin.
* Due to their chemical composition similar to bone tissue, synthetic bone substitutes are an interesting alternative to autografts and allografts which present some inconvenient (quantity to sample, infection of sampling site…).
* Bone substitutes are bioresorbable and replaced by bone during the healing process (bone remodelling).
* Nowadays, bone substitutes represent a common and efficient procedure to treat surgical or traumatic osseous defects. They are indicated and used in various pathologies and types of surgery, but they always have the same intended use: to fill a bone void.
* Bone substitutes are also used in spine surgeries for cage filling and/or posterolateral fusion.

TEKNIMED has developed several bone substitutes currently used in various types of surgery. Due to their increasing use, there is a need of real-life safety and efficacy data on these products.

This retro-prospective study is performed to assess the safety and performance of TEKNIMED bone substitutes in their current clinical use.

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years or older.
* Be willing to sign an informed consent approved by IRB or EC (where applicable) or not being opposed to the use of their clinical data in the study (France) and

  o For prospective inclusion:
* Be considered for a surgery where bone filling with one of the TEKNIMED bone substitutes comprised in this study is needed and intended to be used according to the IFU.

  o For retrospective inclusion:
* Have undergone a surgery with a TEKNIMED bone substitute used according to the IFU, between the 1st January 2015 and the date of the site initiation visit
* Be informed of the study and not being opposed to the use of their clinical data in the study (France) or be willing to sign an informed consent (where applicable) during the first follow-up visit following the site initiation.

Exclusion Criteria:

Patients presenting one of the following conditions will not be included:

* Under trusteeship or guardianship
* Pregnancy or breast-feeding women

According to contraindications per IFU:

* Procedures other than those stated in the INDICATIONS section
* Patients susceptible to allergic reactions to the product components.

CERAFORM®, TRIHA+®:

- Treatment of large bone defects which could impact the stability of bone structure without implementing a mechanical stabilisation system (such as plate(s), screw(s), nail(s), cage(s))

NANOGEL®:

* Use in vertebroplasty procedures
* Subcutaneous use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People presenting a bone defect created by surgical or traumatic injury.
Sampling Method: Non-Probability Sample
Enrollment: 425 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2032-09-30 (Estimated)

PRIMARY OUTCOMES:
Successful bone repair | 24 months
  Evaluated through the rate of revision surgery due to a failure of the substitute.

SECONDARY OUTCOMES:
Alleviation of Pain | 24 months
  Pain evaluated by Visual Analogue Scale (VAS): on a scale of 0 to 10, with 0 being no pain and 10 being the most severe pain at the Baseline and at the Follow-up visits
Bone reconstruction | 24 months
  Evaluated on X-Rays by the Lane and Shadu score and the healing stage
Well-being | 24 months
  Evaluated through a series of short questions : On a scale from 0 (Not at all) to 10 (Perfectly well)
  1. Are you satisfied with your global health status? _____ / 10
  2. Do you manage to carry out your day-to-day activities? _____ / 10
  3. Do you manage to achieve what you would like? _____ / 10
  4. Do you feel relaxed _____ / 10
  5. Do you feel fit / with energy? _____ / 10
  6. Do your physical, psychic and emotional conditions allow you to enjoy your relationships with others? _____ / 10
Patient satisfaction | 24 months
  Evaluated through a series of short questions A. Are you satisfied with your surgery? YES/NO/Without opinion B. Has your health improved? YES/STABLE/NO C. Given the results, would you do this intervention again? YES/NO/Without opinion

CONTACTS AND LOCATIONS:
Locations (6):
- France (5):
  - Pôle Rachis Hôpital Privé d'Eure et Loir, Mainvilliers, Eure et Loir
  - Hôpital Joseph Ducuing, Toulouse, Haute Garonne
  - Clinique Médipole Garonne, Toulouse, Haute Garonne
  - CHRU Brabois, Nancy, Meurthe et Moselle
  - Clinique du Pré, Le Mans, Sarthe
- OCM Klinik GmbH, München, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No